CLINICAL TRIAL: NCT05111678
Title: Neurological Symptoms and Findings in Individuals Exposed to Indoor Air Pollutants
Status: Completed | Type: Observational
Sponsor: Turku University Hospital (Other Government)
Responsible Party: Sponsor
Other Study IDs: 1/2021
Record Dates: First submitted 2021-08-02; First posted 2021-11-08 (Actual); Last update posted 2024-04-10 (Actual); Status verified 2024-04

CONDITIONS: Exposure to Polluted Air

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood and cerebrospinal fluid
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Indoor air pollutant groups: 50 patients that have been exposed to indoor air pollutants
- Neurological symptoms groups: 50 patients with neurological symptoms possibly due to adverse external exposure without any exposure to indoor air pollutants
- Healthy controls: 25 healthy age- and gender-matched controls

SUMMARY:
To evaluate neurological findings with TSPO-PET and MRI in patients who have been exposed to indoor air pollutants and have potentially neurological symptoms.

DETAILED DESCRIPTION:
Health problems related to indoor air pollutants have been studied for several decades but there is still not sufficient scientific evidence to prove the association between many of the described symptoms and exposure to mold and other air pollutants.

This research aims on studying the activation of microglia and inflammation in the brains of individuals exposed to indoor air pollutants having neurological symptoms with MRI and TSPO-PET imaging, questionnaires and biomarkers and compare the findings to individuals having neurological conditions without exposure to indoor air pollutants as well as healthy controls.

ELIGIBILITY:
Inclusion Criteria:

All:

* Signing the informed consent form
* Adults over 18 years of age

Indoor air pollutant groups:

* Exposed to indoor air pollutants
* Neurological symptoms

Neurological symptoms groups:

* Neurological symptoms possibly due to adverse external exposure

Healthy controls:

* Reported healthy person

Exclusion Criteria:

All:

* Pregnancy or breast-feeding
* Corticosteroid treatment within 4 weeks of imaging
* Patients with claustrophobia, or a history of moderate to severe anxiety disorder or panic attacks (which could potentially lead to preterm termination of the imaging)
* Contraindication to PET scan and MRI investigations
* Exposure to experimental radiation in the past 12 months such that radiodosimetry limits would be exceeded by participating in this study.
* Intolerance to previous PET scans; i.e. previous hypersensitivity reactions to any PET ligand or imaging agent or failure to participate in and comply with previous PET scans.

Neurological symptoms groups and healthy controls:

* Exposure to indoor air pollutants

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study will recruit 50 patients who have been exposed to indoor air pollutants and have possibly neurological symptoms. For comparison the study will recruit also 50 patients with neurological symptoms due to a possible adverse external exposure and who have not been exposed to indoor air pollutants. Additionally, 25 healthy controls will be included.
Sampling Method: Non-Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-03-31 (Actual)

PRIMARY OUTCOMES:
[11C]PK11195 binding in the brain | Baseline
  Change in microglial activity in the brains of the individuals in different study groups as measured by [11C]PK11195 PET imaging

SECONDARY OUTCOMES:
DTI-MRI metrics | Baseline
  To evaluate the microstructural damage of the brain between individuals in different groups
Results from questionnaires | Baseline
  Questionnaires about quality of life compared between the indoor air pollutant and neurological symptoms groups
Blood biomarkers | Baseline
  Biomarkers measured from blood to assess the possible inflammatory state of individuals in different study groups
Neurography measures | Baseline
  Done additionally if clinical studies indicate necessary, to assess the state of peripheral nerves
Electromyography measures | Baseline
  Done additionally if clinical studies indicate necessary, rating each examined muscle as normal/myopathic/neuropathic
Cerebrospinal fluid biomarkers | Baseline
  Biomarkers measured from cerebrospinal fluid to assess the possible inflammatory state of individuals in different study groups

CONTACTS AND LOCATIONS:
Overall Officials: Laura Airas, MD,Professor, Principal Investigator — Turku University Hospital, division of clinical neurosciences
Locations (1):
- Turku PET Centre, Turku, Southwest Finland, Finland